CLINICAL TRIAL: NCT02111421
Title: Optimal Dose of Dexmedetomidine Sedation Following Spinal Anesthesia: Postpartum Versus Nonpregnant Women
Brief Title: Postpartum Women's Dexmedetomidine Sedation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Responsible Party: Principal Investigator, bo xu, associate chief physician, Guangzhou General Hospital of Guangzhou Military Command
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cesarean Surgery
Record Dates: First submitted 2014-04-07; First posted 2014-04-11 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Cesarean Section
Keywords: dexmedetomidine; parturient; nonpregnant women; sedation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- parturients (Experimental): Parturients after the umbilical cord was clapped in cesarean section were accepted an initial dose of 1.0 μg/kg dexmedetomidine, with dose adjustment intervals of 0.1μg/kg in first three turning points and 0.05μg/kg in the last four turning points.
  Interventions: Drug: Dexmedetomidine 01
- nonpregnant women (Experimental): Nonpregnant women were accepted an initial dose of 1.0 μg/kg dexmedetomidine, with dose adjustment intervals of 0.1μg/kg in first three turning points and 0.05μg/kg in the last four turning points.
  Interventions: Drug: Dexmetomidine 02

INTERVENTIONS:
Drug: Dexmedetomidine 01 — Initial dose of dexmedetomidine was 1.0 μg/kg, with dose adjustment intervals of 0.1μg/kg in first three turning points and 0.05μg/kg in the last four turning points,after the umbilical cord was clapped.The wight used to calculate the dose of dexmedetomidine would be that the total weight of the mother minus the weight of the placenta, amniotic fluid and fetal.
  Arms: parturients
Drug: Dexmetomidine 02 — Initial dose of dexmedetomidine was 1.0 μg/kg, with dose adjustment intervals of 0.1μg/kg in first three turning points and 0.05μg/kg in the last four turning points,as soon as the spinal anesthesia
  Arms: nonpregnant women

SUMMARY:
Currently, spinal anesthesia is most commonly used for cesarean section.But spinal anesthesia can not block the visceral vagus nerve, and the patients are prone to nausea, vomiting, chest tightness or other discomfort when the uterus is stretched .For parturients who have poor uterine contractions and are bleeding larger, obstetricians often use oxytocin to strengthen the contraction of the uterine,which also would increase the parturients' discomfort.Anesthesiologists often intravenous sedative hypnotics (eg.propofol or midazolam) to alleviate the fear of the parturients after the baby is delivered.One of the side effects of propofol or midazolam is that they would lead to the respiratory depression.For the poor respiratory reserve of the parturients, functional residual capacity(FRC) of this group could be reduced by up to 20%, and the oxygen consumption was also increased.The SPO2 could decline quickly intraoperatively.Dexmedetomidine is a novel , highly selective α2 adrenergic receptor agonists , and its selectivity for α2 receptor is 1600 times higher than α1.It also could provide dose-dependent sedation , analgesia , anti-anxiety and inhibition of sympathetic nerves and other effects.Because of its minimal impact on the respiratory , it could safely and effectively used to sedate patients undergoing cesarean section.But the change of endocrine system and hemodynamic of the parturients may affect the pharmacokinetics and pharmacodynamics of some anesthetic drugs.Currently studies have demonstrated the increased sensitivity of some anesthetic drug in parturients, such as lidocaine and isoflurane.The study is aim to explore the optimal dexmedetomidine dose to produce suitable sedation in parturients ,and compared with norman nonpregnant women.

DETAILED DESCRIPTION:
Parturients undergo cesarean section and normal nonpregnant women undergo lower abdominal surgery were scheduled . All patients accepted spinal anesthesia first.And then an dose of dexmedetomidine would be performed after umbilical cord was clapped in the parturients and in non-pregnant women group the dose of dexmedetomidine would be performed after the spinal anesthesia was conducted.Initial doses was 1.0μg/kg,with dose adjustment intervals of 0.1μg/kg in first three turning points and 0.05μg/kg in the last four turning points. Each patient's sedation state was assessed using the modified observer's assessment of awareness /sedation (OAA/S) scale every 5 min after starting the dexmedetomidine infusion for 30 min. Adequate sedation was defined as an OAA/S≤3 at any assessment time point during the 30 min

ELIGIBILITY:
Inclusion Criteria:

1. ASA Ⅰ ~ Ⅱ women undergoing cesarean surgery under spinal anesthesia
2. ASA Ⅰ ~ Ⅱ nonpregnancy women undergoing lower abdominal surgery under spinal anesthesia
3. Written informed consent from the patient or the relatives of the participating patient
4. nonpregnancy women BMI:18～25 kg/m2 , parturients BMI <35kg/m2

Exclusion Criteria:

1. Mental illness can not match
2. Spinal anesthesia contraindicated
3. People who have Slow-type arrhythmias
4. People who were language or hearing impaired
5. Sensory block reached to T6 or higher.
6. People who had lung infection or sleep apnea syndrome.
7. Chronic renal failure
8. Alcohol or drug abuse
9. Already taking gabapentin, pregabalin, benzodiazepin or antidepression drug

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
The assessment of sedation | every 5 min after starting the dexmedetomidine infusion for 30 min
  The aim of our study is to define the median effective sedative dose (ED50) of dexmedetomidine for providing adequate sedation in cesarean surgery,using the Dixon up-and-down method. Adequate sedation was defined as an OAA/S≤3 at any assessment time point during the 30 min after dexmedetomidine infusion.

SECONDARY OUTCOMES:
comparision of ED50 | every 5 min after starting the dexmedetomidine infusion for 30 min
  compare the ED50 between postpartum parturients and nonpregnant women

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Military Region General Hospital, Department of Anesthesiology, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Xiong M, Chen B, Hu Z, Gupta S, Li Z, Liu J, He J, Patel S, Eloy JD, Xu B. Dose Comparison of Dexmedetomidine Sedation following Spinal Anesthesia: Parturient versus Nonpregnant Women-A Randomized Trial. Anesthesiol Res Pract. 2020 Jul 27;2020:1059807. doi: 10.1155/2020/1059807. eCollection 2020. PMID 32802051